CLINICAL TRIAL: NCT05353153
Title: The Psychological Experience of Pathological Pregnancy. Study of the Case of Premature Rupture of Membranes and Evaluation of the Impact of Hypnosis Support
Acronym: HYPNOPROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Laboratory of Psychopathology and Health Processes, University of Paris (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021_0409; 2021-A02139-32 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Preterm Premature Rupture of Membrane
Keywords: PPROM; hypnosis; psychology; anxiety; complicated pregnancy
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Anxiety Disorders; Pregnancy Complications | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypnosis group (Experimental)
  Interventions: Other: hypnosis
- Control group (Active Comparator)
  Interventions: Other: standart care

INTERVENTIONS:
Other: hypnosis — Hypnosis-based intervention with two sessions of hypnosis (focusing on the treatment of anxiety)
  Arms: hypnosis group
Other: standart care — no intervention no hypnosis
  Arms: Control group

SUMMARY:
This research investigates the impact of a hypnosis-based intervention in alleviating state anxiety in Preterm Premature Rupture of Membranes (PPROM). Our main hypothesis is that a two-session intervention can decrease anxiety for pregnant women with PPROM compared to usual care. This research also studies the impact of the experience of a PPROM during a pregnancy on several variables such as perinatal depression, pregnancy-related anxiety, bonding and childbirth experience, as well as control and pain perceived during chilbirth. Our hypotheses are that the experience of PPROM negatively influences these variables, and that this impact is alleviated by the hypnosis-based intervention for the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Being an adult French-speaking woman,
* primi or multipara,
* less than 33 weeks and 6 days of amenorrhea
* having being diagnosed with PPROM

Exclusion Criteria:

* Women cognitively impaired or with important hearing issues,
* being placed under protective measures,
* caring more than one fetus,
* having a severe, preexisting or triggered during the pregnancy,
* psychiatric pathology,
* caring a fetus with an abnormality having required further medical investigations, or participating in another clinical trial comprising an intervention measuring psychological variables

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — no upper age limit, all women at age to reproduct
Enrollment: 60 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
State anxiety by STAI-Y-A scale | between baseline and 3-week (+/- 1 week) prenatal measurement
  change in anxiety-status level between baseline and 3-week (+/- 1 week) the STAI-Y-A scale, which is a 20-item self-questionnaire evaluating anxiety at the present time. The measurement is done on a Likert scale from 1 to 4 (each number corresponding to a value, 1 being the lowest and 4 the highest for each item, score ranging from 20 to 80).

SECONDARY OUTCOMES:
Pregnancy related anxiety by PRAQ-R2 | 1 time at baseline
  The Pregnancy related Anxiety Questionnaire revised is a 10-item Self-administered questionnaire that assesses specific prenatal anxiety. On a Likert scale ranging from 1 to 5 (each number corresponding to a value, 1 being the lowest and 4 the hghest for each item, score ranging from 10 to 50)
Pregnancy related anxiety by PSAS | At 4 time points: 2 in the prenatal period (at baseline and 3 weeks after) and 2 in the postnatal period (at 1 day to 7 days postpartum and at 4 to 6 weeks postpartum)
  The Postnatal Specific Anxiety Scale (PSAS) is a 44-item self-administered questionnaire that assesses specific postpartum anxiety. On a Likert scale ranging from 1 to 4 (each number corresponding to a value, 1 being the lowest and 4 the highest for each item, score ranging from 44 to 176)
State anxiety by STAI-Y-A | between the baseline measurement and the postnatal measurements ( at 1 day to 7 days postpartum and at 4 to 6 weeks postpartum)
  The change in anxiety-status level between the baseline measurement and the postnatal measurements
Perinatal depression by EPDS | At 3 time points: 2 in the prenatal period (at baseline and 3 weeks after) and 1 in the postnatal period ( at 4 to 6 weeks postpartum)
  the EPDS is a self-administered questionnaire assessing the presence of depressive symptoms in the pre- and postnatal period. This scale has 10 items with a score ranging from 0 to 30, the threshold score is 10.5
Childbirth experience by QEVA | At 1 day to 7 days postpartum
  The french version of the questionnaire for assessing childbirth experience QACE.
  this is a 17 item self-questionnaire evaluating the childbirth experience, with a score ranging from 0 to 51, the highest score being the more negative experience.
Labor agentry by LAS ( Labor Agentry Scale) | at one point at 1day to 7 days postpartum
  this is a 32-item self-administered questionnaire evaluating the perceived control during childbirth. the score tanges from 32 to 210, the highest score evaluating a higher perceived control.
Perinatal bonding by PAI | At one point at baseline
  the Prenatal Attachement Inventory (PAI) is a 21-item self-administered questionnaire assessing bonding in the prenatal period, on a Likert scale ranging from " almost nerver" to almost always", with a total score ranging from 21 to 84, a higher score evaluating a higher bonding
postnatal bonding by PPBQ | at 4 to 6 weeks postpartum
  The Postpartum Bonding Questionnaire (PPBQ) is a 22-item self-administered questionnaire assessing bonding in the postpartum period, on a Likert scale ranging from "always" to "never", with a total score ranging from 0 to 110. A cut-off score of 26 has been indicated as the onset of bonding disorder, and 40 for more severe disorders in bonding with the child
Pain Visual Analog Scale by EVA | At 2 time points in the postnatal period : at 1 day to 7 days postpartum and at 4 to 6 weeks postpartum
  The VAS (Visual Analog Scale) is a self-assessment scale of pain, on a 10cm ruler graduated in mm, ranging from "No pain" to "Maximum pain imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Sara BALAGNY, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez, Had, Chu Lille, Lille, France